CLINICAL TRIAL: NCT00775307
Title: A Randomized, Double-blind, Placebo-controlled Phase II-III Multi-centre Study to Evaluate the Effect of Adjuvant Pazopanib (GW786034) Versus Placebo on Post-surgical Disease-free Survival in Patients With Stage I Non Small Cell Lung Cancer and Tumor Size Equal or Inferior to 5 cm.
Brief Title: Adjuvant Pazopanib in Stage I NSCLC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IFCT-0703; Eudract : 2008-004897-41
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-small cell lung cancer; Stage I; adjuvant therapy; Adjuvant Drug Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pazopanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Placebo Comparator): Placebo 400 mg/day (24 weeks)
  Interventions: Drug: Placebo
- A (Experimental): Pazopanib 400 mg/day (24 weeks)
  Interventions: Drug: PAZOPANIB

INTERVENTIONS:
Drug: PAZOPANIB — 400 mg/day (24 weeks)
  Arms: A
Drug: Placebo — Placebo 400 mg/day (24 weeks)
  Arms: B

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of pazopanib compared with placebo in patients with T < or = 5 cm, N0 (stage I according to TNM 2009) completely resected NSCLC.

DETAILED DESCRIPTION:
The study will be conducted in two phases as follows:

* The Phase II component of the study will be a randomized, double-blind, placebo-controlled, multi-centre study performed in France only. After undergoing NSCLC resection, 140 patients will be randomized to receive either pazopanib 400 mg per day or placebo for 24 weeks.
* The Phase III component of the study will be a randomized, double-blind, placebo-controlled, multi-centre study performed internationally. Patients who have completed the Phase II component of the study will be followed and included in the Phase III. Additional patients will also be recruited to a planned total of 355 patients per treatment arm. New patients will be randomized to receive either pazopanib 400 mg per day or placebo for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Complete resection of the primary tumour and local extension has to be performed. All margins must be free of microscopical disease. At the time of resection, a complete mediastinal lymph-node resection or lymph-node sampling is required. Surgeons are encouraged to dissect or sample all accessible nodal levels.
2. Single surgically resected pathological stage I NSCLC lesion: consisting of a tumor < 5 cm in greatest dimension (see TNM staging on Appendix 10).
3. No regional lymph node involvement.
4. Pre-operative petscan
5. Satisfactory healing of surgical wound.
6. Patients >= 18 and < 70 years of age.
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
8. Recruited to the study and available to start treatment investigational product at least 4 weeks but no longer that 8 weeks after the surgical resection of the NSCLC.
9. No approved or investigational anti-cancer therapy concurrently or in the 5 years prior to start of study drug, including tumor embolization, chemotherapy, radiation therapy, immunotherapy, hormone therapy, biologic therapy, or anti angiogenic therapy (e.g., inhibitors of VEGF or VEGFR).
10. Adequate organ system function
11. Ability to swallow and retain oral medication.
12. 12. A female is eligible to enter and participate in this study if she is of:

    Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has undergone:
    * Hysterectomy.
    * Bilateral oophorectomy (ovariectomy).
    * Bilateral tubal ligation.
    * Or who is post-menopausal:
    * Patients not using hormone replacement therapy (HRT) must have experienced total cessation of menses for ≥1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone value >40 mIU/mL and an estradiol value <40 pg/mL (<140 pmol/L).
    * Subject using HRT must have experienced total cessation of menses for ≥ 1 year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT.

    Childbearing potential, including any female who has had a negative serum pregnancy test within 1 week prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception. Contraceptive methods acceptable to the IFCT, when used consistently and in accordance with both the product label and the instructions of the physician, are as follow:
    * An intrauterine device with a documented failure rate of less than 1% per year.
    * Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry and is the sole sexual partner for that female.
    * Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product.
    * Double-barrier contraception : condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)
    * Oral contraceptive, either combined or progestogen alone [Hatcher, 2004]
    * Injectable progestogen [Hatcher, 2004]
    * Implant of levonorgestrel [Hatcher, 2004]
    * Estrogenic vaginal ring [Hatcher, 2004]
    * Percutaneous contraceptive patches [Hatcher, 2004]

    Female patients who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 15 days following the last dose of study drug.

    A male with a female partner of childbearing potential is eligible to enter and participate in the study if he uses a barrier method of contraception or abstinence during the study.
13. French Patients: in France, a patient will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security insurance.

Exclusion Criteria:

1. Prior malignancy. Note: Patients who have had another malignancy and were treated more than 5 years ago and have since been considered cured, or patients with a history of basocellular skin carcinoma or in situ carcinoma of the uterine cervix are eligible.
2. Presence of any concurrent disease or condition that would make the subject inappropriate for study participation including any unresolved or unstable, serious toxicity from prior administration of another investigational drug or any serious medical disorder that would interfere with the subject's safety, obtaining informed consent, or compliance with all study related procedures.
3. Major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks prior to beginning therapy, or anticipation of the need for a major surgical procedure during the course of the study.
4. History or clinical evidence of nodal or distant metastases (screening of brain metastasis is mandatory).
5. Bronchioalveolar carcinoma of lobar or multi lobar involvement. Bronchioalveolar carcinomas presenting as a discrete solitary radiological mass or nodule are eligible.
6. History of human immunodeficiency virus infection or chronic hepatitis B or C.
7. History of hemoptysis after resection of lung cancer.
8. Clinically significant gastrointestinal anomalies including, but not limited to:

   * Malabsorption syndrome
   * Disease significantly affecting gastrointestinal function or major resection of the stomach or small bowel that could affect the absorption of study drug.
   * Active peptic ulcer disease
   * Inflammatory bowel disease
   * Ulcerative colitis, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis or other gastrointestinal condition increasing the risk of perforation.
   * History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment
9. Presence of active or uncontrolled infection.
10. Evidence of active bleeding or bleeding diathesis.
11. History of any one or more of the following cardiovascular conditions within the past 6 months:

    * Coronary/peripheral artery bypass graft, cardiac angioplasty or stenting.
    * Myocardial infarction.
    * Severe/unstable angina pectoris.
    * Symptomatic peripheral vascular disease, pulmonary embolism or untreated deep venous thrombosis (DVT), cerebrovascular accident or transient ischemic attack.

    Note : Subject with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible

    • Class III or IV congestive heart failure, as defined by the New York Heart Association (Appendix 5).
12. Poorly controlled hypertension (defined as a systolic blood pressure (SBP) of >= 140 mmHg or diastolic blood pressure (DBP) >= 90 mmHg.

    Note: Initiation or adjustment of anti-hypertensive medication(s) is permitted prior to study entry. Blood pressure (BP) must be re-assessed on two occasions separated by at least 5 minutes. The mean SBP/DBP values from both BP assessments must be <140/90 mmHg in order for a subject to be eligible for the study.
13. Following anomalies on ECG : Q wave, ischemia, QT > 480 msec, atrio-ventricular block 2 or 3, atrial fibrillation
14. Therapeutic anticoagulation treatment.
15. Chronic daily treatment with aspirin (≥ 325 mg/day) or non-steroidal anti-inflammatory agents known to inhibit platelet function. Treatment with dipyridamole, ticlopidine, clopidogrel and/or cilostazol is also not allowed.
16. Pregnant or lactating female.
17. Concurrent treatment with an investigational agent or participation in another clinical trial.
18. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2008-11; Primary Completion 2015-12 (Actual); Study Completion 2016-04-18 (Actual)

PRIMARY OUTCOMES:
Phase II component of the study : Feasibility of regime ; Phase III component of the study : disease-free survival (DFS) | month

SECONDARY OUTCOMES:
Overall survival (OS), Detailed assessment of compliance, Incidence and severity of AEs and other safety measures, Reporting profile of AEs of interest during long-term follow-up, Rates of loco-regional and distant recurrences, Quality of Life | month

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin BESSE, Dr, Principal Investigator — Institut Gustave Roussy (IGR); Jean-Charles SORIA, Pr, Study Director — Institut Gustave Roussy (IGR)
Locations (40):
- France (40):
  - Annemasse - CH, Ambilly
  - Béziers - CH, Béziers
  - Bobigny - Hôpital Avicenne, Bobigny
  - Bordeaux - Polyclinique Nord, Bordeaux
  - Boulogne - Ambroise Paré, Boulogne
  - Caen - Centre François Baclesse, Caen
  - Caen - CHU Côte de Nacre, Caen
  - Clamart - Hôpital Percy, Clamart
  - Clermont Ferrand - CHU, Clermont-Ferrand
  - Colmar - CH, Colmar
  - Dax - CH, Dax
  - Grenoble - CHU, Grenoble
  - Le Mans - Centre Hospitalier, Le Mans
  - Lille - Hôpital Calmette, Lille
  - Mantes La Jolie - CH, Mantes-la-Jolie
  - Marseille - Hôpital Sainte Marguerite, Marseille
  - Metz - Clinique Claude Bernard, Metz
  - Mont de Marsan - CH, Mont-de-Marsan
  - Montpellier - Clinique Clémentville, Montpellier
  - Montpellier - CHRU, Montpellier
  - Moulins - CH, Moulins
  - Nantes - Centre René Gauducheau, Nantes
  - Nevers - CH, Nevers
  - CHU, Nîmes
  - Orléans - CH, Orléans
  - Paris - Saint Louis, Paris
  - Paris - hôpital Saint-Antoine, Paris
  - Paris - Hopital Tenon, Paris
  - Pau - CH, Pau
  - Centre Catalan d'Onologie, Perpignan
  - Lyon Sud, Pierre-Bénite
  - Reims - CHU, Reims
  - Rennes - CHU, Rennes
  - Strasbourg - NHC, Strasbourg
  - Thonon les bains - CH, Thonon-les-Bains
  - Toulon - HIA, Toulon
  - Toulouse - CHU Larrey, Toulouse
  - Nancy - CHU, Vandœuvre-lès-Nancy
  - Vesoul - CHI, Vesoul
  - Villejuif - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Besse B, Mazieres J, Ribassin-Majed L, Barlesi F, Bennouna J, Gervais R, Moreau L, Berard H, Debieuvre D, Molinier O, Moro-Sibilot D, Souquet PJ, Jacquot S, Petit L, Lena H, Pignon JP, Lacas B, Morin F, Milleron B, Zalcman G, Soria JC; Intergroupe Francophone de Cancerologie Thoracique (IFCT). Pazopanib or placebo in completely resected stage I NSCLC patients: results of the phase II IFCT-0703 trial. Ann Oncol. 2017 May 1;28(5):1078-1083. doi: 10.1093/annonc/mdx070. PMID 28327934
- See also: IFCT official website — http://www.ifct.fr